CLINICAL TRIAL: NCT06964607
Title: Impact of Sodium Glucose Co-transporter 2-Inhibitors on Clinical Outcome and Left Ventricular Function in Patients Presented by Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Asmaa Atef Hussein Mohammed, Resident of Cardiovascular Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264MS145/4/23
Record Dates: First submitted 2025-04-19; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Sodium-glucose Cotransporter 2; Inhibitors; Clinical Outcome; Left Ventricule; Acute Myocardial Infarction
MeSH Terms: interventions — empagliflozin; dapagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sodium-glucose cotransporter-2 Inhibitors group: Patients received conventional management of acute myocardial infarction and reperfusion therapy as indicated, plus one of the available sodium-glucose co-transporter-2 Inhibitors in Egypt (Empagliflozin or Dapagliflozin), irrespective of the presence or absence of diabetes mellitus or type of heart failure(HFrEF, HFmEF, HFpEF).
  Interventions: Drug: Sodium-glucose cotransporter-2 Inhibitors
- Conventional treatment group: Patients received conventional management of acute myocardial infarction and reperfusion therapy as indicated without adding sodium-glucose co-transporter-2 inhibitors.
  Interventions: Drug: Conventional treatment

INTERVENTIONS:
Drug: Sodium-glucose cotransporter-2 Inhibitors — Patients received conventional management of acute myocardial infarction and reperfusion therapy as indicated, plus one of the available sodium-glucose co-transporter-2 Inhibitors in Egypt (Empagliflozin or Dapagliflozin), irrespective of the presence or absence of diabetes mellitus or type of heart failure(HFrEF, HFmEF, HFpEF).
  Other Names: Empagliflozin or Dapagliflozin
  Groups: Sodium-glucose cotransporter-2 Inhibitors group
Drug: Conventional treatment — Patients received conventional management of acute myocardial infarction and reperfusion therapy as indicated without adding sodium-glucose co-transporter-2 inhibitors.
  Groups: Conventional treatment group

SUMMARY:
This study aimed to assess the effect of adding sodium glucose co-transporter two inhibitors on clinical outcome and left ventricular function in patients with acute myocardial Infarction.

DETAILED DESCRIPTION:
Sodium-glucose co-transporter-2 (SGLT-2) inhibitors are a class of anti-hyperglycemic agents that act on the SGLT-2 proteins expressed in the renal proximal convoluted tubules. They exert their effect by preventing the reabsorption of filtered glucose from the tubular lumen.

Early initiation and continuation of SGLT2 inhibition for acute myocardial infarction is appealing with many proposed mechanistic effects that may alter the natural history, predisposition to ventricular remodeling, and progression to chronic heart failure and end-stage heart disease

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* Recent myocardial infarction.

Evidence of significant myocardial necrosis defined as a rise in troponin level > 99th Percentile ULN (upper limit of normal). In addition, at least one of the following criteria must be met:

* Symptoms of ischemia.
* ECG changes indicative of new ischemia (new ST-T changes or new Left bundle branch block (LBBB))
* Imaging evidence of new regional wall motion abnormality.

  * Estimated Glomerular Filtration Rate (eGFR)> 30 ml/min/1.73 m2.
  * Blood pressure before first drug dosing >110/70 mmHg.

Exclusion Criteria:

* Known allergy to sodium/glucose cotransporter 2 (SGLT2) inhibitors.
* Patients with poor echocardiographic views.
* Hemodynamic instability as defined by intravenous administration of catecholamine.
* >1 episode of severe hypoglycemia within the last 6 months under treatment with insulin or sulfonylurea.
* Pregnant women or females of childbearing age without adequate contraceptive methods.
* Acute symptomatic urinary tract infection (UTI) or genital infection
* Patients currently being treated with any SGLT-2 inhibitor or having received treatment with any SGLT-2 inhibitor within the 4 weeks before the screening visit.
* Patient with a previous myocardial ischemic event or previous heart failure.
* Patients with significant valvular dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a prospective, non-randomized study had been conducted on 80 patients with newly diagnosed acute myocardial infarction presented to cardiovascular medicine department, Tanta university hospital between April 2023 and April 2024.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Assessment of clinical outcome | 6 months following revascularization
  Clinical outcome was studied at 6 months with notification of any adverse clinical events (ACE) during this period: Patients were followed-up for 6 months with documentation of any ACE including new ischemic event, worsening heart failure symptoms, arrhythmia, re-hospitalization or death, that developed during this period then re-classified into a group that did not develop any adverse clinical events and the other that showed ≥ one adverse clinical events to study the impact of different parameters on the incidence of ACE.

SECONDARY OUTCOMES:
Serum creatinine level | 6 months following revascularization
  Serum creatinine level was recorded.
HbA1C level | 6 months following revascularization
  HbA1C level was recorded.
NT-proBNP level | 6 months following revascularization
  NT-proBNP level was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.